CLINICAL TRIAL: NCT02461732
Title: Randomized Controlled Trial of a Novel Cognitive-Behavioral Treatment for Posttraumatic Stress and Substance Dependence
Brief Title: Trial of a Novel Cognitive-Behavioral Treatment for Posttraumatic Stress and Substance Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Anka A Vujanovic, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-14-0486
Record Dates: First submitted 2015-05-22; First posted 2015-06-03 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Posttraumatic Stress Disorder; Substance Dependence
Keywords: posttraumatic stress disorder; PTSD; substance dependence; substance use
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders | interventions — Therapeutics; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT for Substance Dependence (Active Comparator): Standard CBT for substance use disorders
  Interventions: Behavioral: Cognitive-Behavioral Therapy for Substance Dependence
- Integrated CBT for PTSD and Substance Dependence (Experimental): Integrated CBT for PTSD and substance use disorders, combining elements of cognitive processing therapy for PTSD with coping skills and relapse prevention for substance use disorders
  Interventions: Behavioral: Treatment for Integrated Posttraumatic Stress and Substance Use (TIPSS)

INTERVENTIONS:
Behavioral: Treatment for Integrated Posttraumatic Stress and Substance Use (TIPSS) — Topics covered include:
  drug triggers; antecedents/consequences of drug use; relapse prevention; coping skills; problem thinking; changing problem thinking; lifestyle balance; values; increasing non-drug activities; education on PTSD and trauma/PTSD/substance use associations; discussion and written statement of impact of trauma on beliefs about self, others, world; written account of trauma memory and in-session review and discussion; cognitive exercises and cognitive restructuring regarding trauma-related thoughts; review of any between-session trauma-relevant substance use and cravings
  Arms: Integrated CBT for PTSD and Substance Dependence
Behavioral: Cognitive-Behavioral Therapy for Substance Dependence — Topics covered include:
  drug triggers; antecedents/consequences of drug use; relapse prevention; coping skills; problem thinking; changing problem thinking; lifestyle balance; values; increasing non-drug activities
  Arms: CBT for Substance Dependence

SUMMARY:
The purpose of the study is to determine whether a novel integrated cognitive-behavioral treatment for posttraumatic stress disorder (PTSD) and substance dependence (i.e., Treatment for Integrated Posttraumatic Stress and Substance use; TIPSS) is more effective than cognitive-behavioral treatment for substance dependence alone with regard to PTSD symptoms and substance use quantity and frequency.

DETAILED DESCRIPTION:
The proposed study is a randomized controlled clinical trial, comparing the efficacy of two cognitive-behavioral therapy (CBT) interventions: standard CBT for substance dependence and a novel integrated CBT program for PTSD and substance dependence. The study will run for approximately 3 years. A total of 100 participants will be enrolled at a rate of 4 participants per month over 25 months to ensure that 80 participants complete the protocol (presuming 20% attrition). Each participant will attend 12 treatment sessions, meeting twice per week for 6 weeks. Treatment sessions will last 1-hour each.

Primary study outcomes will include frequency and quantity of substance use and PTSD symptom severity. Substance use-related outcomes will include: rates of substance abstinence, as measured by (1) urine toxicology testing, (2) alcohol breath level analyses, and (3) participants' self-report of substance use. PTSD symptom outcomes will include symptom severity ratings as measured by clinical interview (i.e., Clinician-Administered PTSD Scale-5; CAPS-5) and self-report (Posttraumatic Checklist; PCL-5).

Secondary study outcomes will include examination of mediational effects. Specifically, changes in distress tolerance, as indexed via self-report (Distress Tolerance Scale) and computer/behavioral tasks (i.e., Mirror-Tracing Task, Paced Auditory Serial Addition Task-Computerized Version, Breath-Holding Task), are expected during the course of the treatment. Changes in cue reactivity are also expected over the course of treatment, as indexed by decreased psychophysiological reactivity (heart rate, respiration rate) during script-driven imagery tasks (listening to trauma/drug related scripts vs. netural). A total of four sessions (baseline/screening and sessions 4, 8, 12) will be preceded by the laboratory sessions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* English language proficiency
* Current (past month) substance dependence, noting exclusions as delineated below
* History of trauma exposure, as per DSM-5 Criterion A1 definition
* Current (past month) PTSD symptoms: score of at least 25 on PCL-5 and/or at least 4 symptoms of moderate severity (scored 2 or higher) endorsed on CAPS-5
* Seeking treatment for trauma-related symptoms and substance dependence

Exclusion Criteria:

* Exclusive [only] nicotine dependence
* Alcohol dependence requiring detoxification
* Opiate dependence requiring detoxification
* Current or past bipolar I disorder
* Current or past major psychotic disorder
* Active (past 6 months) psychotic spectrum symptoms
* Major unstable medical conditions
* Current (past month) suicidal ideation with intent and/or plan
* Current (past month) homicidal ideation with intent and/or plan
* Inability to provide verbal/written consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
PTSD Symptoms | for the duration of the study / through the conclusion of treatment, up to 8 weeks
  PCL-5 self-report measure: severity of symptoms
Substance Use | for the duration of the study / through the conclusion of treatment, up to 8 weeks
  (1) rates of substance abstinence, as measured via urine toxicology testing, alcohol breath level analyses, and participants' self-reports of substance use; (2) longest sustained abstinence, defined as the maximum number of self-reported days of abstinence for each participant.
PTSD Diagnosis | for the duration of the study / through the conclusion of treatment, up to 8 weeks
  CAPS interview measure: severity of symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Science Center at Houston - Center for Neurobehavioral Research on Addiction, Houston, Texas, United States